CLINICAL TRIAL: NCT02379052
Title: A Randomized, Double-Blind, Parallel, Placebo-Controlled Study of the Efficacy, Safety and Tolerability of Dupilumab in Adult Patients With Active Eosinophilic Esophagitis
Brief Title: Study of Dupilumab in Adult Participants With Active Eosinophilic Esophagitis (EoE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R668-EE-1324
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dupilumab 300 mg QW (Experimental): Participants received SC dupilumab 300 mg during the 12-week double-blind treatment phase. Participants received 2 injections (300-mg initial dose, followed by a 300-mg loading dose) on day 1, followed by weekly injections.
  Interventions: Drug: Dupilumab
- Placebo (Experimental): Participants received matching placebo once weekly (qw) during the 12-week double-blind treatment phase. Participants received 2 injections on day 1, followed by weekly injections.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab
  Other Names: DUPIXENT®; REGN668(SAR231893)
  Arms: Dupilumab 300 mg QW
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to assess the clinical efficacy of repeat subcutaneous (SC) doses of dupilumab, compared with placebo, to relieve symptoms in adult participants with active, moderate to severe Eosinophilic Esophagitis (EoE).

The secondary objectives of the study are:

* To assess the safety, tolerability, and immunogenicity of SC doses of dupilumab in adult participants with active, moderate to severe EoE
* To assess the effect of dupilumab on esophageal eosinophilic infiltration
* To evaluate the pharmacokinetics (PK) of dupilumab in adult participants with EoE

ELIGIBILITY:
Key inclusion criteria:

1. Documented diagnosis of EoE by endoscopy prior to or at screening
2. History of on average at least 2 episodes of dysphagia (with intake of solids off anti-inflammatory therapy) per week in the 4 weeks prior to screening and on average at least 2 episodes of documented dysphagia per week in the weeks between screening and baseline; dysphagia is defined as trouble swallowing solid food, or having solid food stick, by participant report
3. Must remain on a stabilized diet for at least 6 weeks prior to screening and during the course of the study; stable diet is defined as no initiation of single or multiple elimination diets or reintroduction of previously eliminated food groups
4. Documented history of or presence of any of the following: allergic disease (e.g, allergic asthma, allergic rhinitis, atopic dermatitis (AD), or food allergies), peripheral eosinophil counts ≥0.25 GI/L, or serum total Immunoglobulin E (IgE) ≥100 kU/L

Key Exclusion Criteria:

1. Prior participation in a dupilumab (anti-IL-4R) clinical trial
2. Other causes of esophageal eosinophilia or the following diseases: hypereosinophilic syndromes, Churg-Strauss vasculitis, and eosinophilic gastroenteritis
3. History of achalasia, active Helicobacter pylori infection, Crohn's disease, ulcerative colitis, celiac disease, and prior esophageal surgery prior to screening
4. Any esophageal stricture unable to be passed with a standard, diagnostic, adult (9 to10 mm) upper endoscope or any critical esophageal stricture that requires dilation at screening
5. History of bleeding disorders or esophageal varices
6. Use of chronic aspirin, nonsteroidal agents, or anti-coagulants within 2 weeks prior to screening. Participants should not stop these agents solely to become eligible for entry into this study
7. Treatment with an investigational drug within 2 months or within 5 half-lives (if known), whichever is longer, prior to screening
8. Use of systemic corticosteroids within 3 months or swallowed topical corticosteroids within 3 months prior to screening
9. Use of inhaled (pulmonary or nasal) topical corticosteroids within 3 months prior to screening and during the study, except stable dose for at least 3 months prior to screening biopsy, which cannot be changed during the study
10. Treatment with oral immunotherapy (OIT) within 6 months prior to screening
11. Allergen immunotherapy unless on stable dose for at least 1 year prior to screening
12. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study

Note: The list of inclusion/ exclusion criteria provided above is not intended to contain all considerations relevant to a participant's potential participation in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2017-02-17 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (14):
- United States (14):
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Urbana, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Chevy Chase, Maryland
  - Boston, Massachusetts
  - New York, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Salt Lake City, Utah
  - Fairfax, Virginia

REFERENCES:
- [Derived] Wechsler ME, Klion AD, Paggiaro P, Nair P, Staumont-Salle D, Radwan A, Johnson RR, Kapoor U, Khokhar FA, Daizadeh N, Chen Z, Laws E, Ortiz B, Jacob-Nara JA, Mannent LP, Rowe PJ, Deniz Y. Effect of Dupilumab on Blood Eosinophil Counts in Patients With Asthma, Chronic Rhinosinusitis With Nasal Polyps, Atopic Dermatitis, or Eosinophilic Esophagitis. J Allergy Clin Immunol Pract. 2022 Oct;10(10):2695-2709. doi: 10.1016/j.jaip.2022.05.019. Epub 2022 May 28. PMID 35636689
- [Derived] Hamilton JD, Harel S, Swanson BN, Brian W, Chen Z, Rice MS, Amin N, Ardeleanu M, Radin A, Shumel B, Ruddy M, Patel N, Pirozzi G, Mannent L, Graham NMH. Dupilumab suppresses type 2 inflammatory biomarkers across multiple atopic, allergic diseases. Clin Exp Allergy. 2021 Jul;51(7):915-931. doi: 10.1111/cea.13954. Epub 2021 Jun 26. PMID 34037993
- [Derived] Hirano I, Dellon ES, Hamilton JD, Collins MH, Peterson K, Chehade M, Schoepfer AM, Safroneeva E, Rothenberg ME, Falk GW, Assouline-Dayan Y, Zhao Q, Chen Z, Swanson BN, Pirozzi G, Mannent L, Graham NMH, Akinlade B, Stahl N, Yancopoulos GD, Radin A. Efficacy of Dupilumab in a Phase 2 Randomized Trial of Adults With Active Eosinophilic Esophagitis. Gastroenterology. 2020 Jan;158(1):111-122.e10. doi: 10.1053/j.gastro.2019.09.042. Epub 2019 Oct 5. PMID 31593702

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 80 participants were screened, of whom 47 were enrolled at 14 sites. Screen failures did not meet all inclusion criteria, met one or more exclusion criterion, or withdrew consent (33 participants). Of the 47 enrolled, 23 participants were randomized to receive dupilumab 300 mg QW and 24 participants were randomized to receive placebo.
Pre-assignment Details: After providing informed consent, participants were assessed at screening (to occur between day -35 & day -1) for eligibility to participate in the study. Participants who met the eligibility criteria underwent day 1 baseline assessments & randomized in a 1:1 ratio to receive dupilumab or placebo during the 12-week double-blind treatment phase.
Groups:
- Dupilumab 300 mg QW: Participants received subcutaneous (SC) dupilumab 300 mg during the 12-week double-blind treatment phase. Participants received 2 injections (300-mg initial dose, followed by a 300-mg loading dose) on day 1, followed by weekly injections.
Period: Overall Study
Arm/Group | Placebo | Dupilumab 300 mg QW
Started | 24 | 23
Completed | 18 | 18
Not Completed | 6 | 5
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Did Not Meet Inc./ Exclusion Criteria | 1 | 0
Not completed — Subject was Incarcerated | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized patients. Efficacy analyses were based on the treatment allocated by the interactive voice response system (IVRS)/ interactive web response system (IWRS) at randomization (as randomized).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab 300 mg QW | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.1 (12.75) | 33.1 (8.70) | 34.7 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 10 | 13 | 23
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic or Latino | 24 | 23 | 47
Weekly Straumann Dysphagia Instrument (SDI) Patient Reported Outcome (PRO) Score (0-9) [Mean (Standard Deviation); unit: Score on a Scale] — The SDI is a PRO used to determine frequency/ intensity of dysphagia (recall period 1-wk). Frequency of dysphagia events is graded on a 5-pt scale: 0=none, 1=1x/wk, 2=several/wk, 3=1x/day, 4=several/day; intensity is graded on a 6-pt scale: 0=swallowing unrestricted, 1=slight sensation of resistance, 2=slight retching with delay, 3=short period of obstruction necessitating intervention, 4=longer-lasting period of obstruction removable by vomiting, 5=long-lasting complete obstruction requiring endoscopic intervention. Total score ranges from 0-9 (higher score indicates worsening symptoms).
  Score on a Scale | 6.4 (1.01) | 6.4 (1.04) | 6.4 (1.01)
Weekly Reported Eosinophilic Esophagitis Activity Index (EEsAI) PRO Score (0-100) [Mean (Standard Deviation); unit: Score on a Scale] — The EEsAI PRO questionnaire includes items related to the intensity and frequency of dysphagia, the influence of specific food groups on dysphagia symptoms, and other symptoms independent of eating or drinking (ie, heartburn, acid regurgitation, and chest pain). The total EEsAI PRO score ranges from 0 to 100 (higher score indicates worsening symptoms). The EEsAI PRO utilizes 24-hour and
  1-week recall periods. Population: Includes number of participants evaluable for this characteristic
  Score on a Scale
    number analyzed (Participants) | 22 | 23 | 45
    (all) | 62.2 (16.45) | 62.0 (18.36) | 62.1 (17.25)
Adult Eosinophilic Esophagitis Quality of Life (EoE-QOL-A) Total Mean Score (1-5) [Mean (Standard Deviation); unit: Score on a Scale] — The EoE-QOL-A questionnaire includes 30 items related to 5 established domains (eating/diet impact, social impact, emotional impact, disease anxiety, and swallowing anxiety) of daily life experiences. The EoE-QOL-A has a 1-week recall period. The items are graded on a 5-point scale: 1 (Not at All), 2 (Slightly), 3 (Moderately), 4 (Quite a bit), and 5 (Extremely). The EoE-QOL-A score is the average obtained by dividing the total score by the number of questions (for participants without disease, 120/30 = 4). Total scores range from 1 to 5 (higher scores indicate worsening symptoms).
  Score on a Scale | 3.11 (0.995) | 3.02 (0.899) | 3.06 (0.940)
Eosinophilic Esophagitis-Endoscopic Reference Score (EoE-EREFS) Total Score (0-8) [Mean (Standard Deviation); unit: Score on a Scale] — The EoE-EREFS includes a total of 6 major items related to the presence/ severity of esophageal features. Specific features scored by the investigator include rings (absent[0], mild[1], moderate[2], severe[3], not applicable); stricture (yes[1], no[0], not applicable); diameter of the stricture (if applicable; measurement not scored); exudates (absent[0], mild [1], severe[2]); furrows (absent[0], present[1]); edema (absent[0], present[1]). The total score of the 5 scored items ranges from 0 to 8 (higher score indicates worsening symptoms).
  Score on a Scale | 4.3 (1.46) | 3.9 (1.87) | 4.1 (1.67)
Baseline Blood Peripheral Eosinophils (EOS) [Mean (Standard Deviation); unit: Giga/Liter (L)] | 0.43 (0.285) | 0.31 (0.177) | 0.37 (0.242)
Number of Esophageal Dilations [Mean (Standard Deviation); unit: Count of Esophageal Dilations] — Population: Analysis included only participants with any dilations
  Count of Esophageal Dilations
    number analyzed (Participants) | 10 | 11 | 21
    (all) | 3.9 (3.31) | 5.7 (8.03) | 4.9 (6.17)
Age Group [Number; unit: Count of Participants]
  ≥18 to <40 years | 15 | 16 | 31
  ≥40 to <65 years | 9 | 7 | 16
  ≥65 years | 0 | 0 | 0
Baseline Blood Peripheral Eosinophils (EOS) [Number; unit: Count of Participants]
  Number of participants with EOS < 0.25 Giga/L | 8 | 11 | 19
  Number of participants with EOS ≥ 0.25 Giga/L | 16 | 12 | 28
Peak Eosinophils/ High Power Field (eos/hpf) Count [Mean (Standard Deviation); unit: Count of Eosinophils] — Peak eos/hpf was determined by counting eosinophils in the most inflamed areas of each esophageal region sampled at each time point and calculating the change in the peak count at each site.
  Count of Eosinophils | 101.1 (57.12) | 102.1 (53.46) | 101.6 (54.76)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Straumann Dysphagia Instrument (SDI) Patient Reported Outcome (PRO) Total Score at Week 10
Description: The SDI is a PRO used to determine frequency/ intensity of dysphagia (recall period 1-wk). Frequency of dysphagia events is graded on a 5-pt scale: 0=none, 1=1x/wk, 2=several/wk, 3=1x/day, 4=several/day; intensity is graded on a 6-pt scale: 0=swallowing unrestricted, 1=slight sensation of resistance, 2=slight retching with delay, 3=short period of obstruction necessitating intervention, 4=longer-lasting period of obstruction removable by vomiting, 5=long-lasting complete obstruction requiring endoscopic intervention. Total score ranges from 0-9 (higher score indicates worsening symptoms).
Time Frame: Baseline, Week 10
Population: Full Analysis Set (FAS) included all randomized participants. Efficacy analyses were based on the treatment allocated by the interactive voice and web response system (IVRS/IWRS) at randomization (as randomized).
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Score on a Scale | -1.3 (0.57) | -3.0 (0.53)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p = 0.0304, ANCOVA; A 2-step multiple imputation (MI) method addressed missing values ([seeds = 12345 & 54321 in the 2 steps respectively; number of imputations=50]); Least Squares (LS) Mean Difference = -1.7, 95% CI 2-sided [-3.22 to -0.16] — The confidence interval (CI) with p-value is based on treatment difference (dupilumab vs. placebo) of the LS mean using analysis of covariance (ANCOVA) model with baseline measurement as covariate and the treatment as fixed factor

2. Secondary Outcome: Percent Change From Baseline in Straumann Dysphagia Instrument (SDI) Patient Reported Outcome (PRO) Total Score at Week 10
Description: as for outcome 1
Time Frame: Baseline, Week 10
Population: Full analysis set (FAS) included all randomized participants. Efficacy analyses were based on the treatment allocated by the IVRS/IWRS at randomization (as randomized).
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Percent Change | -18.59 (8.978) | -45.05 (8.435)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p = 0.0312, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -26.45, 95% CI 2-sided [-50.523 to -2.387] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Absolute Change From Baseline in Straumann Dysphagia Instrument (SDI) Patient Reported Outcome (PRO) Total Score at Week 12
Description: The SDI is a PRO used to determine frequency/intensity of dysphagia (recall period 1-wk). Frequency of dysphagia events is graded on a 5-pt scale: 0=none, 1=1x/wk, 2=several/wk, 3=1x/day, 4=several/day; intensity is graded on a 6-pt scale: 0=swallowing unrestricted, 1=slight sensation of resistance, 2=slight retching with delay, 3=short period of obstruction necessitating intervention, 4=longer-lasting period of obstruction removable by vomiting, 5=long-lasting complete obstruction requiring endoscopic intervention. Total score ranges from 0-9 (higher score indicates worsening symptoms).
Time Frame: Baseline, Week 12
Population: FAS included all randomized participants. Efficacy analyses were based on the treatment allocated by the IVRS/IWRS at randomization (as randomized).
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Score on a Scale | -2.2 (0.69) | -2.9 (0.56)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p = 0.3830, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-2.48 to 0.96] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percent Change From Baseline in Straumann Dysphagia Instrument (SDI) Patient Reported Outcome (PRO) Total Score at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Percent Change | -31.83 (10.674) | -42.83 (8.573)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p = 0.4147, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -11.00, 95% CI 2-sided [-37.460 to 15.467] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants Achieving a Reduction of ≥ 3 Points in Straumann Dysphagia Instrument (SDI) Patient Reported Outcome (PRO) Total Score From Baseline at Week 10
Description: as for outcome 1
Time Frame: Baseline, Week 10
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Percentage of Participants | 12.5 | 39.1
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p = 0.0490, Clopper-Pearson Exact; Percent Difference = 26.6, 95% CI 2-sided [-3.04 to 51.05] — Difference is Dupilumab minus Placebo. CI = Confidence interval calculated using Clopper-Pearson Exact method

6. Secondary Outcome: Percentage of Participants Achieving a Reduction of ≥ 3 Points in Straumann Dysphagia Instrument (SDI) Patient Reported Outcome (PRO) Total Score From Baseline at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Percentage of Participants | 12.5 | 39.1
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p = 0.0490, Clopper-Pearson Exact; Percent Difference = 26.6, 95% CI 2-sided [-3.04 to 51.05] — Difference is Dupilumab minus Placebo. CI = Confidence interval calculated using Clopper-Pearson Exact method

7. Secondary Outcome: Percent Change From Baseline in Weekly Reported Eosinophilic Esophagitis Activity Index (EEsAI) Patient Reported Outcome (PRO) Score at Week 10
Description: The EEsAI PRO questionnaire includes items related to the intensity and frequency of dysphagia, the influence of specific food groups on dysphagia symptoms, and other symptoms independent of eating or drinking (ie, heartburn, acid regurgitation, and chest pain). The total EEsAI PRO score ranges from 0 to 100 (higher score indicates worsening symptoms). The EEsAI PRO utilizes 24-hour and 1-week recall periods.
Time Frame: Baseline, Week 10
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Percent Change | -11.33 (9.915) | -34.56 (9.076)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p = 0.0850, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -23.23, 95% CI 2-sided [-49.677 to 3.212] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Absolute Change From Baseline in Weekly Reported Eosinophilic Esophagitis Activity Index (EEsAI) Patient Reported Outcome (PRO) Score at Week 10
Description: as for outcome 7
Time Frame: Baseline, Week 10
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Score on a Scale | -9.0 (5.58) | -22.9 (5.01)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p = 0.0635, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -13.9, 95% CI 2-sided [-28.54 to 0.78] — The confidence interval (CI) with p-value is based on treatment difference (dupilumab vs. placebo) of the LS mean using ANCOVA model with baseline measurement and baseline SDI score as covariates and the treatment as fixed factor

9. Secondary Outcome: Percent Change From Baseline in Weekly Reported Eosinophilic Esophagitis Activity Index (EEsAI) Patient Reported Outcome (PRO) Score at Week 12
Description: as for outcome 7
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Percent Change | -3.34 (12.701) | -36.99 (11.168)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p = 0.0608, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -33.65, 95% CI 2-sided [-68.828 to 1.536] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Absolute Change From Baseline in Weekly Reported Eosinophilic Esophagitis Activity Index (EEsAI) Patient Reported Outcome (PRO) Score at Week 12
Description: as for outcome 7
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Score on a Scale | -5.0 (7.06) | -26.1 (5.87)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p = 0.0318, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -21.1, 95% CI 2-sided [-40.42 to -1.86] — [estimate comment as in outcome 8, analysis 1]

11. Secondary Outcome: Percentage of Participants Achieving ≥ 40% Improvement in Weekly Reported Eosinophilic Esophagitis Activity Index (EEsAI) Patient Reported Outcome (PRO) Score From Baseline at Week 10
Description: as for outcome 7
Time Frame: Baseline, Week 10
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Percentage of Participants | 8.3 | 26.1
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p = 0.1365, Clopper-Pearson Exact — P-values were derived by Fisher exact test; CI = Confidence interval calculated using Exact method; Percent Difference = 17.8, 95% CI 2-sided [-11.54 to 43.55] — Difference is Dupilumab minus Placebo

12. Secondary Outcome: Percentage of Participants Achieving ≥ 40% Improvement in Weekly Reported Eosinophilic Esophagitis Activity Index (EEsAI) Patient Reported Outcome (PRO) Score From Baseline at Week 12
Description: as for outcome 7
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Percentage of Participants | 4.2 | 39.1
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p = 0.0044, Clopper-Pearson Exact — P-values were derived by Fisher exact test; CI = Confidence interval calculated using Exact method; Percent Difference = 35.0, 95% CI 2-sided [5.69 to 58.34] — Difference is Dupilumab minus Placebo

13. Secondary Outcome: Percent Change From Baseline in Peak Esophageal Intraepithelial Eosinophils of 3 Esophageal Regions at Week 12
Description: Peak eosinophils/high power field (eos/hpf) was determined by counting eosinophils in the most inflamed areas of each esophageal region sampled at each time point and calculating the change in the peak count at each site.
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Percent Change | 14.23 (12.495) | -92.90 (12.068)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -107.13, 95% CI 2-sided [-141.215 to -73.046] — [estimate comment as in outcome 8, analysis 1]

14. Secondary Outcome: Absolute Change From Baseline in Eosinophilic Esophagitis-Endoscopic Reference Score (EoE-EREFS) by Feature at Week 12
Description: The EoE-EREFS includes a total of 6 major items related to the presence/ severity of esophageal features. Specific features scored by the investigator include rings (absent[0], mild[1], moderate[2], severe[3], not applicable); stricture (yes[1], no[0], not applicable); diameter of the stricture (if applicable; measurement not scored); exudates (absent[0], mild [1], severe[2]); furrows (absent[0], present[1]); edema (absent[0], present[1]). The total score of the 5 scored items ranges from 0 to 8 (higher score indicates worsening symptoms).
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Score on a Scale | -0.3 (0.33) | -1.9 (0.32)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p = 0.0006, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = -1.6, 95% CI 2-sided [-2.50 to -0.68] — [estimate comment as in outcome 8, analysis 1]

15. Secondary Outcome: Change From Baseline in Adult Eosinophilic Esophagitis Quality of Life Questionnaire (EoE-QOL-A) Score at Week 12
Description: The EoE-QOL-A questionnaire includes 30 items related to 5 established domains (eating/diet impact, social impact, emotional impact, disease anxiety, and swallowing anxiety) of daily life experiences. The EoE-QOL-A has a 1-week recall period. The items are graded on a 5-point scale: 1 (Not at All), 2 (Slightly), 3 (Moderately), 4 (Quite a bit), and 5 (Extremely). The EoE-QOL-A score is the average obtained by dividing the total score by the number of questions (for participants without disease, 120/30 = 4). Total scores range from 1 to 5 (higher scores indicate worsening symptoms).
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Score on a Scale | 0.47 (0.141) | 0.80 (0.137)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Test type: Superiority; p = 0.0910, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.33, 95% CI 2-sided [-0.053 to 0.720] — [estimate comment as in outcome 8, analysis 1]

16. Secondary Outcome: Percentage of Participants With Use of Rescue Medication or Procedure (e.g., Esophageal Dilation) Through Week 12
Time Frame: Baseline through Week 12
Population: as for outcome 3
Measure: Number; unit: Percent of Participants
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Percent of Participants | 0 | 0

17. Secondary Outcome: Percent of Participants With Treatment-Emergent Adverse Events (TEAEs) During the Study
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) that developed or worsened or became serious during the on-treatment period (time from the first dose of study drug up to the end of study (Week 28). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-participant hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Baseline through Week 28
Population: The safety analysis set (SAF) included all randomized participants who received any study drug, and were analyzed as treated.
Measure: Number; unit: Percent of Participants
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 24 | 23
Percent of Participants | 66.7 | 91.3

ADVERSE EVENTS:
Time Frame: Adverse event (AE) information was collected from the time the informed consent was signed until the participant's last study visit. Serious adverse event (SAE) information was collected until the event was considered chronic and/or stable.
Description: An AE is any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease which was temporally associated with the use of a study drug, whether or not considered related to the study drug.
  The safety analysis set (SAF) included all randomized participants who received any study drug, and the analyses were based on as treated. The safety analyses were based on the SAF.
Arm/Group | Placebo | Dupilumab 300 mg QW
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 3/23
Other Adverse Events (participants affected / at risk) | 14/24 | 18/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Dupilumab 300 mg QW (N=23)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Dupilumab 300 mg QW (N=23)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (3)
Injection site erythema (General disorders) | 2 (3) | 8 (29)
Injection site inflammation (General disorders) | 0 (0) | 3 (9)
Injection site pain (General disorders) | 2 (3) | 2 (8)
Injection site rash (General disorders) | 0 (0) | 3 (10)
Injection site urticaria (General disorders) | 0 (0) | 2 (10)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (3)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (5)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT02379052/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT02379052/SAP_001.pdf